CLINICAL TRIAL: NCT03607825
Title: ExtracorPoreal FILtration of Subarachnoid Hemorrhage Via SpinaL CAtheteR EXTension
Brief Title: FILtration of Subarachnoid Hemorrhage Via SpinaL CAtheteR Extension
Acronym: PILLAR-XT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnetronix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1.0 11July18
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2021-06

CONDITIONS: Subarachnoid Hemorrhage
Keywords: aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neurapheresis System (Experimental): CSF filtration
  Interventions: Device: Neurapheresis System

INTERVENTIONS:
Device: Neurapheresis System — CSF filtration system and lumbar catheter

SUMMARY:
The objective of this study is to further demonstrate safety and characterize effectiveness of the Neurapheresis™ System (extracorporeal system and catheter) to remove red blood cells (RBCs) and lysed blood by-products from hemorrhagic cerebrospinal fluid (CSF) following aneurysmal subarachnoid hemorrhage (aSAH).

DETAILED DESCRIPTION:
The PILLAR-XT study is designed to further confirm safety and characterize efficacy of Neurapheresis therapy. The study works in tandem with the current SOC treatments for SAH and does not detract from the established care pathways, or deny enrolled subjects proven therapies. The PILLAR-XT study utilizes the established skill sets of chosen Investigators who are already trained in the treatment and care of SAH patients and insertion/management of lumbar drains.

ELIGIBILITY:
Inclusion Criteria:

* Modified Fisher Grade 2, 3 or 4
* Hunt & Hess I-IV
* First aneurysmal SAH
* Patient is ≤ 48 hours post bleeding event
* World Federation of Neurosurgeons (WFNS) Grades I-IV

Exclusion Criteria:

* Pregnancy
* Patients with a SAH due to mycotic aneurysm or AV malformation
* Patients who present with an acute MI or unstable angina
* Imaging demonstrates supratentorial mass lesions > or = 15 cc
* Imaging demonstrates > or = 2 mm of mid-line-shift associated with infarction and or edema
* Effacement of the basilar cisterns
* Vasospasm on admission as defined by angiographic evidence
* Patients with a coagulopathy that cannot be reversed
* Thrombocytopenia def. platelet count < 100,000
* Patients on low molecular weight heparin such as Lovenox
* Non-communicating Obstructive hydrocephalus
* Existing hardware that prevents accurate CT imaging
* Pre-existing Lumbar Drain
* Local skin infections or eruptions over the puncture site
* Signs of CNS systemic infection, sepsis or pneumonia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai, New York, New York
  - Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects were consented but catheter placement was not attempted as they were determined to no longer meet inclusion criteria after they were consented (n=4 Intent to Treat) and were immediately withdrawn. Two subjects were consented and the catheter placement was attempted but was not successful (n=2 Attempt to Treat) and were withdrawn after 2-day follow-up. The remaining subjects (N=27) had successful catheter placement, had CSF Filtration and were followed for 30 days per the protocol.
Period: Overall Study
Arm/Group | Neurapheresis System
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neurapheresis System
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  years
    number analyzed (Participants) | 29
    (all) | 49.9 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  Participants
    number analyzed (Participants) | 29
    Female | 22
    Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 33
Height [Mean (Full Range); unit: cm] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  cm
    number analyzed (Participants) | 29
    (all) | 166.7 [149.9 to 200]
Weight [Mean (Full Range); unit: kg] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  kg
    number analyzed (Participants) | 29
    (all) | 76.1 [46.7 to 125]
History of Smoking [Count of Participants; unit: Participants] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  Participants
    number analyzed (Participants) | 29
    (all) | 16
History of Hypertension [Count of Participants; unit: Participants] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  Participants
    number analyzed (Participants) | 29
    (all) | 18
Prior History of Brain Injury Treatment [Count of Participants; unit: Participants] — Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  Participants
    number analyzed (Participants) | 29
    (all) | 2
WFNS Grading System [Median (Full Range); unit: Units on a Scale] — The WFNS (World Federation of Neurological Surgeons) Grading System For Subarachnoid Hemorrhage combines the Glasgow Coma Scale in the presence (+) or absence (-) of Motor Deficit to create a 1-5 Grade:
  GCS 15, Motor Deficit+ = WFNS Grade 1 GCS 13-14, Motor Deficit- = WFNS Grade 2 GCS 13-14, Motor Deficit+ = WFNS Grade 3 GCS 7-12, Motor Deficit + or - = WFNS Grade 4 GCS 3-6, Motor Deficit + or - = WFNS Grade 5
  A higher WFNS grade (e.g. WFNS Grade 5) is associated with higher mortality rates / worse outcomes. Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  Units on a Scale
    number analyzed (Participants) | 29
    (all) | 2 [1 to 4]
Hunt & Hess Scale [Median (Full Range); unit: units on a scale] — The Hunt and Hess (H&H) Scale is a clinical grading system of subarachnoid hemorrhage that ranges from 1 to 5.
  H&H 1: Asymptomatic, mild headache, slight nuchal rigidity H&H 2: Moderate to severe headache, nuchal rigidity, no neurologic deficit other than cranial nerve palsy H&H 3: Drowsiness/confusion, mild focal neurologic deficit H&H 4: Stupor, moderate-sever hemiparesis H&H 5: Coma, decerebrate posturing Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  units on a scale
    number analyzed (Participants) | 29
    (all) | 3 [1 to 4]
Glasgow Coma Scale [Median (Full Range); unit: units on a scale] — The Glasgow Coma Scale (GCS) is used to describe the level of consciousness after a brain injury. It combines scores of 3 activities: Eye Opening, Motor Response, and Verbal Response. Eye Opening is scored from 1-4, Motor Response from 1-6, and Verbal Response from 1-5. The minimum GCS score is 3 and the maximum is 15.
  For example, a severe brain injury is GCS 8 or less, Moderate is GCS 9-12, and Mild is GCS 13-15 Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  units on a scale
    number analyzed (Participants) | 29
    (all) | 14 [7 to 15]
Modified Fisher Grade [Median (Full Range); unit: units on a scale] — The modified Fisher Grade Scale (mFS) in a means of stating the severity of an aneurysmal subarachnoid hemorrhage based on the amount and type of blood as measured on CT. The scale ranges from 0-4.
  mFS = 0: No SAH, or IVH mFS = 1: Thin diffuse or focal SAH, no IVH mFS = 2: Thin diffuse or local SAH, with IVH mFS = 3: Thick focal or diffuse SAH, no IVH mFS = 4: Thick local or diffuse SAH with IVH Population: In this protocol there were 4 intent to treat patients. Per protocol, the intent to treat patients were not included in this measure
  units on a scale
    number analyzed (Participants) | 29
    (all) | 3 [3 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cisternal Blood From Enrollment to Catheter Removal
Description: Mean Change in Cisternal Blood measured by the Hijdra Score as Documented by CT, represented as a percent change. The Hijdra Score evaluates 10 cisterns and fissures within the brain for the quantity of blood present on a 0-3 scale. 0 means no blood present, 1 is a small amount, 2 is moderately filled, and 3 is completely filled. The 10 scores are added up. A Hijdra Score of 0 means no blood present (normal) and a Hijdra Score of 30 means all the cisterns and fissures are completely filled with blood (poor outcome).
Time Frame: Enrollment to Catheter Removal (Immediately post treatment)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Neurapheresis System
Number analyzed (Participants) | 26
percent change | -64.7 (19.8)

2. Secondary Outcome: Mean Change in Red Blood Cells From Before to After the Treatment Period.
Description: Mean Change in Red Blood Cells as measured by CSF analysis of RBCs, represented as a percent change. The RBCs are measured in the CSF in quantity of RBC (10^6) per mm^3. The change is calculated using the first available RBC measurement (at either Catheter Insertion or after 1 hour of CSF Filtration, if first measurement unavailable) compared to the last available RBC measurement before the catheter was removed.
Time Frame: Catheter Insertion to Catheter Removal (Immediately post treatment)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Neurapheresis System
Number analyzed (Participants) | 26
percent change | -85.8 (20.8)

3. Secondary Outcome: Mean Change in Total Protein From Before to After the Treatment Period
Description: Mean Change in Total Protein as measured by CSF analysis of RBCs, represented as a percent change. The Total Protein is measured in the CSF in quantity of mg/dL. The change is calculated using the first available Total Protein measurement (at either Catheter Insertion or after 1 hour of CSF Filtration, if first measurement unavailable) compared to the last available Total Protein measurement before the catheter was removed.
Time Frame: Catheter Insertion to Catheter Removal (Immediately post treatment)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Neurapheresis System
Number analyzed (Participants) | 26
percent change | -82.4 (16.1)

ADVERSE EVENTS:
Time Frame: enrollment through 30 day follow-up
Description: PILLAR-XT did not track all-cause AEs or AEs related to SOC or the SAH clinical pathway e.g., re-bleed, deep vein thrombosis, skin breakdown etc. Study required event reporting is limited to AEs directly related to the investigational catheter, investigational system or Neurapheresis procedure, or study required element (such as CSF sampling). In cases where the event may have an attributable dual causality the center should report the event.
Arm/Group | Neurapheresis System
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurapheresis System (N=29)
Diencephalic Herniation (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurapheresis System (N=29)
Headache (Nervous system disorders) | 2 (2)
Back Pain (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that first publication of the results of the Study shall be made in conjunction with the presentation of a joint multi-center publication. PI may publish individually if multi-center publication is published, or no multi-center publication is published within 12 months of conclusion, or Sponsor confirms in writing there will be no multi-center publication. If no multi-center publication within 12 months, Sponsor will provide PI access to aggregate data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT03607825/Prot_SAP_000.pdf